CLINICAL TRIAL: NCT01909141
Title: Combined Letrozole-metformin-pioglitazone Versus Combined Clomiphene Citrate-metformin-pioglitazone in Clomiphene Citrate-resistant Women With Polycystic Ovary Syndrome
Brief Title: Ovulation Induction in Women With Clomiphene Citrate Resistant PCOS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Abdel Fattah, lecturer of Obstetrics and Gynecology-Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: fem2013
Record Dates: First submitted 2013-07-15; First posted 2013-07-26 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-09

CONDITIONS: Polycystic Ovary Syndrome; Infertility
Keywords: letrozole; clomiphene citrate; pioglitazone; metformin; ovulation induction; PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility | interventions — Body Mass Index; Luteinizing Hormone; Thyrotropin; Testosterone; Blood Urea Nitrogen

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- arm 1:letrozole-pioglitazone -metformin group (Active Comparator): Arm 1 will receive letrozole 2.5 mg/day starting from the 3rd day of the cycle and for 5 days and (combined pioglitazone 15 mg+ metformin 850 mg) once daily from the first day of the cycle for 10 days.
  Interventions: Drug: induction of ovulation using letrozole-pioglitazone-metformin; Radiation: transvaginal ultrasound; Other: body mass index (BMI) calculation; Other: day 3: follicle stimulating hormone (FSH), luteinizing hormone (LH), thyroid stimulating hormone (TSH), total testosterone; Other: pretreatment blood urea and serum creatinine; Other: serum estradiol (E2) on day 12; Other: serum progesterone on day 21; Other: blood urea and serum creatinine every month
- arm 2: clomiphene citrate-pioglitazone-metformin (Active Comparator): Arm 2 will receive clomiphene citrate 100 mg/day starting from the 3rd day of the cycle for 5 days and (combined pioglitazone 15 mg + metformin 850 mg) once daily from the first day of the cycle for 10 days.
  Interventions: Drug: induction of ovulation using clomiphene citrate-pioglitazone-metformin; Radiation: transvaginal ultrasound; Other: body mass index (BMI) calculation; Other: day 3: follicle stimulating hormone (FSH), luteinizing hormone (LH), thyroid stimulating hormone (TSH), total testosterone; Other: pretreatment blood urea and serum creatinine; Other: serum estradiol (E2) on day 12; Other: serum progesterone on day 21; Other: blood urea and serum creatinine every month

INTERVENTIONS:
Drug: induction of ovulation using letrozole-pioglitazone-metformin — induction of ovulation will be done for arm 1 for 3 consecutive cycles unless pregnancy occured.
  Arms: arm 1:letrozole-pioglitazone -metformin group
Drug: induction of ovulation using clomiphene citrate-pioglitazone-metformin — induction of ovulation for arm 2 will be done in 3 consecutive cycles unless pregnancy occured.
  Arms: arm 2: clomiphene citrate-pioglitazone-metformin
Radiation: transvaginal ultrasound — transvaginal ultrasound will be done starting from day 10 and every 48 hours until finding a follicle of > 18 mm or till day 20 of the cycle
Other: body mass index (BMI) calculation — BMI will be calculated for all women by dividing the weight in kilograms by the height in meters squared
Other: day 3: follicle stimulating hormone (FSH), luteinizing hormone (LH), thyroid stimulating hormone (TSH), total testosterone — baseline hormonal assay (day 3 FSH, LH, TSH and total testosterone) will be done for all women.
Other: pretreatment blood urea and serum creatinine — blood urea and serum creatinine will be assayed before stating induction of ovulation to have baseline levels.
Other: serum estradiol (E2) on day 12 — serum E2 will be assayed on day 12 of the cycle for all women.
Other: serum progesterone on day 21 — serum progesterone will be assayed on day 21 for all women to monitor ovulation.
Other: blood urea and serum creatinine every month — blood urea and serum creatinine will be assayed every month during the treatment period to find out any hazards on kidney functions

SUMMARY:
Polycystic ovary syndrome (PCOS) affects 5-10% of women in childbearing age. Hyperinsulinemia contributes to chronic anovulation commonly encountered in women with PCOS. The first choice therapy is clomiphene citrate (CC). In CC resistant cases, the American College of Obstetrics and Gynecology (ACOG) recommends the use of insulin sensitizer metformin. Other insulin sensitizing agents include rosiglitazone and pioglitazone. Pioglitazone is said to improve fertility and ovulation in patients with PCOS.CC may be associated with poor endometrial thickening due to its antiestrogenic effect. Letrozole may improve this condition. In this study we will compare the effect of combined letrozole-metformin-pioglitazone with that of combined CC-metformin-pioglitazone in ovulation induction in CC-resistant PCOS women.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) affects 5-10% of women in childbearing age. Hyperinsulinemia contributes to chronic anovulation commonly encountered in women with PCOS. The first choice therapy is clomiphene citrate (CC). In CC resistant cases, the ACOG recommends the use of insulin sensitizer metformin. Other insulin sensitizing agents include rosiglitazone and pioglitazone. Pioglitazone is said to improve fertility and ovulation in patients with PCOS.CC has a long half-life (2 weeks), and this may have a negative effect on the cervical mucus and endometrium, leading to discrepancy between ovulation and conception rates. There has been a search for a compound capable of inducing ovulation but devoid of the adverse antiestrogenic effects of CC. recent studies have suggested that letrozole, an aromatase inhibitor, does not possess the adverse antiestrogenic effects of CC and is associated with higher pregnancy rates than CC treatment in patients with PCOS.

In this study we shall compare the effect of combined letrozole-metformin-pioglitazone with that of combined CC-metformin-pioglitazone in ovulation induction in CC-resistant PCOS women.This will be a prospective comparative clinical trial in which 2 groups of women will be generated (groups A and B) using the sealed envelopes randomization method.Group A (40 women) will receive: letrozole 2.5 mg/day from 3rd day of the cycle for 5 days and (pioglitazone 15 mg + metformin 850 mg) once daily from 1st day of the cycle for 10 days. Group B (40 women) will receive clomiphene citrate 100 mg/day from 3rd day of the cycle for 5 days and (pioglitazone 15 mg + metformin 850 mg) once daily from 1st day of the cycle for 10 days. Ovulation will be monitored by vaginal ultrasound and serum estrogen and progesterone.

ELIGIBILITY:
Inclusion Criteria:

* 20-40 years old
* PCOS infertile women resistant to CC for3 cycles

Exclusion Criteria:

* presence of medical disorders as diabetes, hypertension, cardiac problems, liver or kidney diseases, hyperprolactinemia or thyroid dysfunction.
* use of gonadotropins before
* previous ovarian drilling
* presence of urinary symptoms especially bloody urine

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2013-08; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Abdel Fattah Abdel Moety, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- [Derived] El-khayat W, Abdel Moety G, Al Mohammady M, Hamed D. A randomized controlled trial of clomifene citrate, metformin, and pioglitazone versus letrozole, metformin, and pioglitazone for clomifene-citrate-resistant polycystic ovary syndrome. Int J Gynaecol Obstet. 2016 Feb;132(2):206-9. doi: 10.1016/j.ijgo.2015.06.063. Epub 2015 Nov 6. PMID 26613820

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1:Letrozole-pioglitazone -Metformin Group: Arm 1 received letrozole 2.5 mg/day starting from the 3rd day of the cycle and for 5 days and (combined pioglitazone 15 mg+ metformin 850 mg) once daily from the first day of the cycle for 10 days.
  induction of ovulation using letrozole-pioglitazone-metformin: induction of ovulation was done for arm 1 for 3 consecutive cycles unless pregnancy occurred.
  transvaginal ultrasound: transvaginal ultrasound will be done starting from day 10 and every 48 hours until finding a follicle of > 18 mm or till day 20 of the cycle
  body mass index (BMI) calculation: BMI was calculated.
  day 3: follicle stimulating hormone (FSH), luteinizing hormone (LH), thyroid stimulating hormone (TSH), total testosterone: baseline hormonal assay (day 3 FSH, LH, TSH and total testosterone) were done for all women.
  serum estradiol (E2) was done on day of hCG administration for all women.
  serum progesterone on day 21 was done for all women.
- Arm 2: Clomiphene Citrate-pioglitazone-metformin: Arm 2 received clomiphene citrate 100 mg/day starting from the 3rd day of the cycle for 5 days and (combined pioglitazone 15 mg + metformin 850 mg) once daily from the first day of the cycle for 10 days.
  induction of ovulation using clomiphene citrate-pioglitazone-metformin: induction of ovulation for arm 2 was done in 3 consecutive cycles unless pregnancy occurred.
  transvaginal ultrasound: transvaginal ultrasound was done starting from day 10 and every 48 hours until finding a follicle of > 18 mm or till day 20 of the cycle
  body mass index (BMI) calculation: BMI was calculated.
  day 3: follicle stimulating hormone (FSH), luteinizing hormone (LH), thyroid stimulating hormone (TSH), total testosterone: baseline hormonal assay (day 3 FSH, LH, TSH and total testosterone) were done for all women.
  serum estradiol (E2) was done on day of hCG administration for all women.
  serum progesterone on day 21 was done for all women.
Period: Overall Study
Arm/Group | Arm 1:Letrozole-pioglitazone -Metformin Group | Arm 2: Clomiphene Citrate-pioglitazone-metformin
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1:Letrozole-pioglitazone -Metformin Group: Arm 1 received letrozole 2.5 mg/day starting from the 3rd day of the cycle and for 5 days and (combined pioglitazone 15 mg+ metformin 850 mg) once daily from the first day of the cycle for 10 days.
  induction of ovulation using letrozole-pioglitazone-metformin: induction of ovulation was done for arm 1 for 3 consecutive cycles unless pregnancy occurred.
  transvaginal ultrasound: transvaginal ultrasound was done starting from day 10 and every 48 hours until finding a follicle of > 18 mm or till day 20 of the cycle
  body mass index (BMI) calculation: BMI was calculated.
  day 3: follicle stimulating hormone (FSH), luteinizing hormone (LH), thyroid stimulating hormone (TSH), total testosterone: baseline hormonal assay (day 3 FSH, LH, TSH and total testosterone) were done for all women.
  serum estradiol (E2) was done on day of hCG administration for all women.
  serum progesterone on day 21 was done for all women.
- Arm 2: Clomiphene Citrate-pioglitazone-metformin: Arm 2 will received clomiphene citrate 100 mg/day starting from the 3rd day of the cycle for 5 days and (combined pioglitazone 15 mg + metformin 850 mg) once daily from the first day of the cycle for 10 days.
  induction of ovulation using clomiphene citrate-pioglitazone-metformin: induction of ovulation for arm 2 was done in 3 consecutive cycles unless pregnancy occured.
  transvaginal ultrasound: transvaginal ultrasound was done starting from day 10 and every 48 hours until finding a follicle of > 18 mm or till day 20 of the cycle
  body mass index (BMI) calculation: BMI was calculated.
  day 3: follicle stimulating hormone (FSH), luteinizing hormone (LH), thyroid stimulating hormone (TSH), total testosterone: baseline hormonal assay (day 3 FSH, LH, TSH and total testosterone) were done for all women.
  serum estradiol (E2) was done on day of hCG administration for all women.
  serum progesterone on day 21 was done for all women.
- Total: Total of all reporting groups
Arm/Group | Arm 1:Letrozole-pioglitazone -Metformin Group | Arm 2: Clomiphene Citrate-pioglitazone-metformin | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.8 (3.62) | 26.58 (2.9) | 26.19 (3.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Egypt | 50 | 50 | 100
infertility period [Mean (Standard Deviation); unit: years] | 2.67 (1.62) | 3.07 (1.46) | 2.87 (1.5)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.45 (2.84) | 26.57 (2.7) | 26.51 (2.75)
waist/hip ratio [Mean (Standard Deviation); unit: ratio] | 0.838 (0.02) | 0.837 (0.04) | 0.837 (0.037)
systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 106.08 (8.81) | 107.04 (8.97) | 106.56 (8.86)
diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 69.6 (5.31) | 68.44 (5.89) | 69.02 (5.61)
hirsutism [Number; unit: participants] | 11 | 10 | 21
acne [Number; unit: participants] | 7 | 4 | 11
ovarian volume [Mean (Standard Deviation); unit: ml] | 14.17 (0.76) | 14.58 (1.42) | 14.19 (0.98)
FSH [Mean (Standard Deviation); unit: mIU/L] | 5.71 (1.34) | 5.68 (1.38) | 5.7 (1.35)
LH [Mean (Standard Deviation); unit: mIU/L] | 9.81 (3.16) | 10.55 (3.25) | 10.18 (3.21)
E2 [Mean (Standard Deviation); unit: Pmol/dL] | 49.83 (7.31) | 47.75 (10.02) | 48.24 (8.56)
prolactin [Mean (Standard Deviation); unit: ng/ml] | 15.52 (4.84) | 14.3 (5.6) | 14.9 (5.24)
total testosterone [Mean (Standard Deviation); unit: nmol/L] | 1.19 (0.25) | 1.13 (0.2) | 1.16 (0.23)
free testosterone [Mean (Standard Deviation); unit: Pmol/dL] | 3.87 (0.61) | 4.12 (1.17) | 3.99 (0.94)
TSH [Mean (Standard Deviation); unit: mIU/L] | 3.42 (0.61) | 3.51 (0.44) | 3.47 (0.53)
free T4 [Mean (Standard Deviation); unit: nmol/L] | 13.78 (0.84) | 13.58 (0.45) | 13.68 (0.68)

OUTCOME MEASURES:

1. Primary Outcome: Ovulation Rate
Time Frame: 3 months
Measure: Number; unit: percentage of all cycles
Groups:
- Arm 1:Letrozole-pioglitazone -Metformin Group: Arm 1 receivde letrozole 2.5 mg/day starting from the 3rd day of the cycle and for 5 days and (combined pioglitazone 15 mg+ metformin 850 mg) once daily from the first day of the cycle for 10 days.
  induction of ovulation using letrozole-pioglitazone-metformin: induction of ovulation was be done for arm 1 for 3 consecutive cycles unless pregnancy occured.
  transvaginal ultrasound: transvaginal ultrasound was done starting from day 10 and every 48 hours until finding a follicle of > 18 mm or till day 20 of the cycle
  body mass index (BMI) calculation: BMI was caculated.
  day 3: follicle stimulating hormone (FSH), luteinizing hormone (LH), thyroid stimulating hormone (TSH), total testosterone: baseline hormonal assay (day 3 FSH, LH, TSH and total testosterone) were done for all women.
  serum estradiol (E2) was done on day of hCG administration for all women.
  serum progesterone on day 21 was done for all women.
- Arm 2: Clomiphene Citrate-pioglitazone-metformin: Arm 2 received clomiphene citrate 100 mg/day starting from the 3rd day of the cycle for 5 days and (combined pioglitazone 15 mg + metformin 850 mg) once daily from the first day of the cycle for 10 days.
  induction of ovulation using clomiphene citrate-pioglitazone-metformin: induction of ovulation for arm 2 was done in 3 consecutive cycles unless pregnancy occured.
  transvaginal ultrasound: transvaginal ultrasound was done starting from day 10 and every 48 hours until finding a follicle of > 18 mm or till day 20 of the cycle
  body mass index (BMI) calculation: BMI was calculated
  day 3: follicle stimulating hormone (FSH), luteinizing hormone (LH), thyroid stimulating hormone (TSH), total testosterone: baseline hormonal assay (day 3 FSH, LH, TSH and total testosterone) were done for all women.
  serum estradiol (E2) was done on day of hCG administration for all women.
  serum progesterone on day 21 was done for all women.
Arm/Group | Arm 1:Letrozole-pioglitazone -Metformin Group | Arm 2: Clomiphene Citrate-pioglitazone-metformin
Number analyzed (Participants) | 50 | 50
percentage of all cycles | 93 | 108

2. Secondary Outcome: Number of Follicles>18mm.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: follicles
Arm/Group | Arm 1:Letrozole-pioglitazone -Metformin Group | Arm 2: Clomiphene Citrate-pioglitazone-metformin
Number analyzed (Participants) | 50 | 50
follicles | 1.44 (0.16) | 1.5 (0.86)

3. Secondary Outcome: Endometrial Thickness
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Arm 1:Letrozole-pioglitazone -Metformin Group | Arm 2: Clomiphene Citrate-pioglitazone-metformin
Number analyzed (Participants) | 50 | 50
mm | 10.56 (1.79) | 9.68 (1.39)

4. Secondary Outcome: Pregnancy Rate
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Arm 1:Letrozole-pioglitazone -Metformin Group | Arm 2: Clomiphene Citrate-pioglitazone-metformin
Number analyzed (Participants) | 50 | 50
participants | 28 | 24

5. Other Pre Specified Outcome: Safety of Pioglitazone as Regards Serum Creatinine
Description: serum creatinine was measured at the end of the study period (after 3 months) in both groups.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm 1:Letrozole-pioglitazone -Metformin Group | Arm 2: Clomiphene Citrate-pioglitazone-metformin
Number analyzed (Participants) | 50 | 50
mg/dL | 0.62 (0.04) | 0.57 (0.03)

ADVERSE EVENTS:
Arm/Group | Arm 1:Letrozole-pioglitazone -Metformin Group | Arm 2: Clomiphene Citrate-pioglitazone-metformin
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes